CLINICAL TRIAL: NCT00782847
Title: A Prospective Controlled Randomized Multicenter Trial to Evaluate the Effect of a Structurized Multifactorial Behavior Modifying Consultation and Support Programme DiaNe for People With Diabetic Nephropathy
Brief Title: Evaluation Study for the Programme DiaNe for People With Diabetic Nephropathy
Acronym: DiaNe
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: DiaNe HCM GmbH (Other)
Collaborators: Roche Pharma Deutschland GmbH, Grenzach-Wyhlen, Germany (Unknown); Institute for Medical Outcom Research GmbH, Loerrach, Germany (Unknown)
Responsible Party: Ludwig Merker, MD, Diabetes- und Nierenzentrum Dormagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DiaNe-Studie
Record Dates: First submitted 2008-10-30; First posted 2008-10-31 (Estimated); Last update posted 2008-10-31 (Estimated); Status verified 2008-10

CONDITIONS: Diabetic Nephropathy
Keywords: diabetes mellitus; diabetic nephropathy; hypertension
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- with DiaNe program (Active Comparator): study subjects which participated in the DiaNe consultation and support program
  Interventions: Behavioral: DiaNe consultation and support program
- without DiaNe program (No Intervention): study subjects which received standard care by diabetologist and/or nephrologist

INTERVENTIONS:
Behavioral: DiaNe consultation and support program — the DiaNe consultation and support program for clients with diabetic nephropathy consists of 4 sessions at 90-120 minutes conducted every week in a period of 4 weeks
  Other Names: DiaNe program, DiaNe(R)
  Arms: with DiaNe program

SUMMARY:
This study is designated to evaluate the effect of a patients' educational program called DiaNe® for consultation and support people with diabetic kidney disease in an early stage. The aim of the study is to examine if the program is suitable to stop deterioration of kidney function and to maintain or improve glycemic control. The consultation and support program DiaNe® substantially contributes to a better understanding of the affected clients for this complex clinical picture, allows them for specific interventions and creates the rationale for an active therapeutic relationship.

DETAILED DESCRIPTION:
According to statistics diabetes mellitus is considered to be the leading cause for end stage renal disease in Germany, approximately 35% of the patients starting on dialysis are affected by diabetes-induced nephropathy. This can be seen in countries all over the world. This situation has been known for years. To date, neither structured intervention methods nor educational programs have been designed for and targeting those affected, which would consequently allow for structured, multifactorial intervention at an early stage of diabetic nephropathy. Multifactorial interventions, as published in the Steno-2 trial, appear to be highly effective with regard to long-term complications of diabetes. In order to realize this approach for the affected as well as the medical staff caring for patients with diabetes-induced nephropathy we developed DiaNe®, a consultation and support program, which is designed to give detailed information to the affected in order to induce behavioral changes. We were able to show a clinically significant reduction of microalbuminuria within a first monocenter evaluation trial. We wanted to verify this effect by means of a prospective multicenter randomized cohort trial according to GCP-ICH guidelines.

ELIGIBILITY:
Inclusion Criteria:

* diabetes mellitus
* proven diabetic nephropathy by histological/lab findings and/or discretion of nephrologist
* ability to understand the German language

Exclusion Criteria:

* end stage renal disease and/or dialysis
* unable or unwilling to follow the protocol
* pregnant women
* discretion of nephrologist

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2004-07; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
deterioration of kidney function in diabetic nephropathy | 13 months

SECONDARY OUTCOMES:
HbA1c | 13 months

CONTACTS AND LOCATIONS:
Overall Officials: Ludwig F Merker, MD, Principal Investigator — Diabetes- und Nierenzentrum Dormagen
Locations (1):
- Diabetes- und Nierenzentrum Dormagen, Dormagen, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Cashmore BA, Cooper TE, Evangelidis NM, Green SC, Lopez-Vargas P, Tunnicliffe DJ. Education programmes for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 Aug 22;8(8):CD007374. doi: 10.1002/14651858.CD007374.pub3. PMID 39171639